CLINICAL TRIAL: NCT05417399
Title: Ecological Validity of Clinical Gait Analysis in Children With Cerebral Palsy: Influence of the Hawthorne Effect and Dual-tasks. A Pilot Study
Brief Title: Influence of Hawthorne Effect and Dual-tasks on Gait in CP
Status: Recruiting | Type: Observational
Sponsor: Roessingh Research and Development (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-13822
Record Dates: First submitted 2022-06-09; First posted 2022-06-14 (Actual); Last update posted 2024-05-01 (Actual); Status verified 2024-04

CONDITIONS: Cerebral Palsy; Gait Disorders, Neurologic; Hawthorne Effect; Dual-tasks; Kinematics
MeSH Terms: conditions — Cerebral Palsy; Gait Disorders, Neurologic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
It is the clinical experience of the authors that some children with cerebral palsy who walk in crouch gait show sufficient knee extension during the clinical gait analysis, but walk in considerable knee flexion when they leave the gait laboratory. Possible differences between walking in a gait lab and walking in daily life may be caused by the effect of observational awareness in the lab (also known as the Hawthorne effect), and the lack of dual-tasks (DT) during the analysis (which are common during daily life walking). Since so far there is no technique to reliably measure gait kinematics in children with CP outside of the laboratory, the researchers aim to objectify the influence of both the Hawthorne effect and dual-tasks by introducing different conditions during a standard clinical 3D gait analysis.

DETAILED DESCRIPTION:
Study design: Observational study

Study population: Patients with cerebral palsy, bilateral spastic, knee flexion gait pattern, GMFCS classification I-III, age 4-16 years.

Objective: To determine the effect of observational awareness (the Hawthorne effect) and dual-tasks on spatiotemporal and kinematic variables during a clinical 3D gait analysis.

Primary research question:

Does reduced observational awareness and/or introduction of a dual-task influence knee flexion in stance phase in children with spastic diplegie cerebral palsy and knee flexion gait?

Secondary research questions:

1. Does reduced observational awareness and/or introduction of a dual-task increase toe walking in children with spastic diplegie cerebral palsy and knee flexion gait?
2. In children with spastic diplegic cerebral palsy and knee flexion gait, do spatiotemporal gait parameters change when observational awareness is reduced and/or a dual-task is introduced?

Conditions in which gait data will be gathered:

1. With awareness of observation + without Dual-task
2. With awareness of observation + with Dual-task
3. Without awareness of observation + without Dual-task
4. Without awareness of observation + with Dual-task

ELIGIBILITY:
Inclusion Criteria:

* Cerebral palsy, bilateral spastic, GMFCS classification I-III
* Age <16 years
* Use of bilateral AFO's (rigid or ground reaction AFO's) to improve knee extension in stance

Exclusion Criteria:

* Behavioural issues or poor instructability which might affect participation in the protocol
* Significant visual disorders
* Other diagnoses influencing gait
* Not willing to sign informed consent before inclusion

Ages: 4 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All subjects are recruited from the patient base of Roessingh Center for Rehabilitation. Subjects will be included in the study when a clinical 3D gait analysis is due and the inclusion and exclusion criteria as mentioned are met.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Minimal knee flexion during the single support phase | Day 1
  Minimal knee flexion during the single support phase

SECONDARY OUTCOMES:
Foot to floor angle at initial contact | Day 1
Knee flexion at initial contact | Day 1
Foot to floor angle at moment of minimal knee flexion in single support phase | Day 1
Variation of knee kinematics in stance phase | Day 1
  Calculated with the Winters-Waveform Coefficient of variation
Variation of ankle kinematics in stance phase | Day 1
  Calculated with the Winters-Waveform Coefficient of variation
Walking speed | Day 1
Cadence | Day 1
Step length | Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Hans Rietman, Professor, Study Chair — Roessingh Research and Development
Locations (1):
- Roessingh Research and Development, Enschede, Overijssel, Netherlands

IPD SHARING:
Plan to Share IPD: No